CLINICAL TRIAL: NCT03756844
Title: Effectiveness of the Just Right Challenge Food Club for Decreasing Food Selectivity and Increasing Mealtime Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Michelle A Suarez, PhD, OTRL, Associate Professor, Western Michigan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JRCFC Single-Subject
Record Dates: First submitted 2018-11-12; First posted 2018-11-28 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Food Selectivity
Keywords: Avoidant Restrictive Food Intake Disorder
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Intervention Model Description: This was a single-subject (time series design).
Masking Description: There was no masking. This was a single subject study. Participants allowed us to use their clinical data for research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Just Right Challenge Food Club Protocol (Experimental): There was only one arm in this study. All participants received the Just Right Challenge Food Club Protocol and single subject (time series) data was collected.
  Interventions: Behavioral: Just Right Challenge Food Club

INTERVENTIONS:
Behavioral: Just Right Challenge Food Club — Systematic desensitization, positive reinforcement and escape extinction at a level of just right challenge.

SUMMARY:
This single subject study tested the effectiveness of the Just Right Challenge Food Club for decreasing food selectivity and increasing mealtime qualify for children with developmental disabilities.

DETAILED DESCRIPTION:
This study used a single subject design to test the effectiveness of the Just Right Challenge Food Club for decreasing food selectivity and increasing mealtime quality for children with developmental disabilities. Baseline data was collected during the time that participants spent on the wait list for treatment. Treatment data was collected each week during treatment session. This protocol produced a significant change in both the number of foods the children in the study ate as well as the parents perception of mealtime quality.

ELIGIBILITY:
Inclusion Criteria:

* Children who accepted less than 15 foods as part of their regular diet
* Children who refused whole food groups

Exclusion Criteria:

* Children with life threatening food selectivity per parent report and physician referral information

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Food Inventory questionnaire | Every week for up to 45 weeks
  Parents marked the foods that their child ate over the past week every week for up to 45 weeks

SECONDARY OUTCOMES:
Change in About Your Child's Eating questionnaire | Up to 45 weeks between pre and post test measures.
  A measure of parent perception of mealtime qualify

IPD SHARING:
Plan to Share IPD: No